CLINICAL TRIAL: NCT00438334
Title: Real-World Benefit From Directional Microphone Hearing Aids
Brief Title: Real-World Benefit From Directional Hearing Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 000170
Record Dates: First submitted 2006-12-05; First posted 2007-02-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Hearing Loss
Keywords: Benefit; Directional microphones; Hearing; Hearing aids; Hearing loss; Noise; Objective benefit; Signal-to-noise ratio; Speech understanding; Subjective benefit
MeSH Terms: conditions — Hearing Loss

INTERVENTIONS:
Device: Programmable directional/omni-directional hearing aid

SUMMARY:
Directional microphone hearing aids have been shown to provide benefit for individuals with hearing loss in a number of laboratory experiments. However, few studies have investigated the real-world, subject-reported benefit from these hearing aids, and even fewer have examined directional hearing aid benefit across varying degrees of hearing loss. This study will summarize data from a three-year, multi-faceted study of directional hearing aid benefit. Ninety four subjects were divided into three hearing loss groups (normal-to-moderate, mild-to-moderately-severe, and moderate-to-profound). These subjects were then fit with experimental hearing aids set to either directional or omnidirectional mode to determine if significant differences were present in hearing aid outcomes (both subjective and objective). Both subject and experimenter were blinded to the hearing aid settings. Following one month of use in each experimental setting, subjects completed: probe microphone measurements, speech understanding in noise testing, use questionnaires, subjective benefit scales, and satisfaction scales. At the conclusion of the study, subjects rated their preferences for the experimental settings in quiet, noise and overall. Both objective measures, as well as subjective data, were analyzed across hearing aid and hearing loss conditions.

DETAILED DESCRIPTION:
Subjects- 105 subjects were recruited for participation in this study, thirty-five in each of three hearing loss groups. Subjects were assigned to the three groups according to the severity of their hearing losses. Group 1 (mild) subjects exhibited normal sloping to moderately severe SNHL, with Pure Tone Averages (PTAs) at 500, 1000, and 2000 Hz of less than 35 dB HL. Group 2 (moderate) consisted of subjects with mild sloping to moderately severe SNHL with PTAs of 35 to 50 dB HL. Group 3 (severe) subjects exhibited moderately-severe, sloping to severe-profound SNHL, with PTAs of greater than 50. All subjects had sloping hearing loss defined as at least a 20 dB average difference between 3000 Hz and 500 Hz. (Due to subject drop-out, the final data consisted of 32 subjects in the mild group, 33 in moderate group, and 29 in the severe group)

Hearing status was assessed by means of audiometric pure-tone and speech recognition testing in a group of previous hearing aid users. Normal middle ear function was verified by means of immittance measures. All subjects exhibited absence of significant air-bone gap at any frequency (<10 dB) and normal tympanograms defined as compensated static admittance between 0.25 and 2.5 mmho measured from the positive tail with tympanometric peak pressure between -150 and +100 daPa. All subjects were service-connected veterans who are eligible for care and amplification through the VA Audiology service. All subjects were previous wearers of binaural hearing aids, with a minimum daily usage requirement of 4 hours/day. All subjects were previous users of output compression hearing aids from the same manufacturer.

All subjects participated in approximately eight to ten hours of testing over the course of four visits. At the first visit, subjects received a hearing test, unaided speech understanding in noise measures, and aided speech understanding in noise with their current hearing aids. Additionally, earmold impressions were obtained for the experimental hearing aids. At the second visit, subjects completed the first set of subjective measures for the unaided and current (own) hearing aid conditions. Subjects were then fit with digitally programmable user-selectable directional/omnidirectional hearing aids in the first of two experimental settings (randomly selected between directional/omnidirectional and omnidirectional only), which they used for approximately one month before returning for the next test session. At the third visit, subjects again completed the entire test battery for the experimental hearing aid worn during the last month. The experimental hearing aid was then programmed for the other condition (directional/omnidirectional or omnidirectional only). At the fourth and final visit, subjects completed the entire test battery for this final hearing aid condition. Additionally, at the final visit, subjects completed a preference questionnaire.

Speech understanding in noise tests:

The Connected Sentence Test (CST) and the Hearing In Noise Test (HINT) were administered to all subjects. An investigator in the room with the subject scored the test. The investigator was blinded to the experimental settings of the hearing aids to control for experimenter bias. The CST is a test of speech intelligibility for everyday speech presented at a fixed SNR. The test consisted of 24 pairs of speech passages produced conversationally. The subject's task was to repeat all words of each test sentence. Each passage included 25 key words that were scored correct or incorrect. Subject scores from 1 pair of passages were averaged to obtain an intelligibility score for each experimental condition. Data from Pearsons et al. indicate that real-world SNRs in relatively noisy environments range from approximately +4 dB to -1 dB. Consequently, the tests were administered at a +3 dB SNR, which represented a relatively difficult real-world listening situation. This SNR was chosen to minimize floor and ceiling effects for all subject groups based on a previous investigation in our laboratory, given the steep performance-intensity function that has been reported for the CST.

The HINT was administered as a second test of sentence intelligibility in noise. For this investigation, two blocks of ten sentences were used for each condition. Listeners were required to repeat sentences spoken by a male talker in the presence of a speech-shaped noise, which was presented at a fixed level of 65 dBA. The level of the speech stimuli was adjusted adaptively until a Speech Reception Threshold (SRT) was determined. The SRT was defined as the SNR necessary for a listener to recognize the speech materials correctly 50 % of the time. Correct identification of each sentence was based on proper repetition of all words of the sentence, with minor exceptions. These exceptions related to the fact that small substitutions in verb tense and the articles "a" and "the" were allowed without scoring a sentence as incorrect. Presentation level of the sentences was adjusted based on the subjects' responses (an incorrect response raised the level; a correct response lowered the level for the next sentence). The level was varied in 4 dB steps for the first 5 trials, and 2 dB steps for the final 15 trials.

Speech in noise test environment:

The arrangement of the speakers for the speech-in-noise testing is shown in figure 1. Both of the speech-in-noise tests were administered in a conference room (5.05 X 4.71 X 2.60 meters) with moderate reverberation (average reverberation time Rt60: 482 ms, measured for octave frequencies from 250 through 4000 Hz, under experimental conditions with 2 people in the room). Each subject was seated in the center of the room with an eight-speaker configuration for the presentation of the speech and noise stimuli. Speech will be presented from a point-source loudspeaker (Tannoy System 600, fused-concentric driver) at a 0º azimuth. Uncorrelated noise was delivered from the seven bipolar loudspeakers (Definitive Technologies BP-2X) spaced equally about the listener [approximately 25, 76, 128, 180, 232, 284, 335]. The use of bipolar loudspeakers allowed for a more diffuse source position in comparison to standard, front-firing loudspeakers. All speakers were equidistant (1.5m) from the subject's head. Speech and noise levels were controlled using a Pentium IV class computer and an eight-channel level controller (Ashly VCM-88).

Hearing aid fitting protocol:

Hearing aid gain was determined using the National Acoustics Laboratory-Revised (NAL-R) prescriptive targets and verified using real-ear (Fonix 6500) measurements. Hearing aid frequency-gain parameters were adjusted so that the measured real ear aided response matched the target response as closely as possible for octave frequencies from 500 to 4000 Hz for both omnidirectional and directional modes. The matches to target are reported in the results. The processing strategy of the experimental hearing aids was set as output compression to match each subject's previous hearing aids. Targets were matched for a 65 dB SPL composite noise input. A real ear saturation response was obtained with a 90 dB SPL broadband input to ensure that high-level stimuli did not exceed listener discomfort levels, and the hearing aid output was adjusted accordingly. In order to maintain a double-blind experiment, the hearing aid programming, fitting, and real ear measurements were performed by one investigator who recorded how the hearing aid was set (omnidirectional or directional) for each visit. This investigator kept these data until the subject completed all aspects of the study. Furthermore, the investigator who programmed and fit the hearing aids was not involved in further data collection with that subject.

Since all subjects were previous users of binaural amplification, a brief orientation to the use of the experimental hearing aids should be sufficient. Subjects were issued a remote control with a volume control and three program buttons. Program 1 was set with the default setting (directional or omnidirectional). In order to ensure subject safety, an omnidirectional program was included in program two across both conditions; however, subjects were instructed only to use program two in situations where it was necessary to hear sounds from all angles equally (e.g. crossing the street in traffic, etc.). Program three on the remote control was set to mute, so that subjects could use only the first two programs. Subjects were be given identical instructions for both settings (omnidirectional and directional) and the investigator who gave the instructions did not know which setting was currently in the subject's hearing aids. Subjects were told that the hearing aids are likely to work best in noise if they could position themselves so that the signal of interest is in front of them and the interfering noise behind. Subjects were instructed on cleaning, care, battery usage, and volume control adjustment. Subjects were asked to wear the experimental hearing aids as much as possible during waking hours, minimally 6 hours/day. Subjects were asked to log their daily hearing aid use on a log sheet that will be provided to verify that they met the 6 hour/day. Additionally, subjects recorded how much time each day was spent in each of the two programs.

Subjective measures:

PHAB- The investigator who administered the subjective measures was masked as to the experimental settings of the hearing aids. All subjects completed the Profile of Hearing Aid Benefit (PHAB) questionnaire for each condition: unaided, previous aid, experimental directional, and experimental omnidirectional. The PHAB is a 66-item inventory that was developed for research usage to generate a measure of hearing aid benefit. Subjects completed the 66 items once for unaided listening and once for each aided condition. The test instrument was scored based on the benefit provided for aided versus unaided conditions.

SADL- All subjects completed the Satisfaction with Amplification in Daily Living (SADL) questionnaire for each of the three aided conditions. The SADL was designed to quantify satisfaction with hearing aids. This scale consists of 15 items in four subscales: positive effects of amplification, service and costs, negative features, and personal image. Subjects respond to questions about their general opinions of wearing hearing aids. For the current study, the 3 questions on cost and service were omitted, because the subjects did not pay for the hearing aids, only wore the experimental hearing aids for one month before completing the survey.

Preference questionnaire- At the conclusion of a subject's involvement in the study, he/she was asked which hearing aid was preferred for quiet and noisy environments as well as if she/he had an overall preference for any of the three hearing aid conditions.

ELIGIBILITY:
Inclusion Criteria:

* 105 subjects were recruited for participation in this study, thirty-five in each of three hearing loss groups.
* Subjects were assigned to the three groups according to the severity of their hearing losses.
* Group 1 (mild) subjects exhibited normal sloping to moderately severe SNHL, with Pure Tone Averages (PTAs) at 500, 1000, and 2000 Hz of less than 35 dB HL.
* Group 2 (moderate) consisted of subjects with mild sloping to moderately severe SNHL with PTAs of 35 to 50 dB HL.
* Group 3 (severe) subjects exhibited moderately-severe, sloping to severe-profound SNHL, with PTAs of greater than 50.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-04; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Probe microphone measurements
Speech understanding in noise
Hearing aid use time
Hearing aid benefit
Hearing aid preference
Hearing aid satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: David Gnewikow, Ph.D., Principal Investigator — Vanderbilt University
Locations (1):
- Department of Veterans Affairs Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Gnewikow D, Ricketts T, Bratt GW, Mutchler LC. Real-world benefit from directional microphone hearing aids. J Rehabil Res Dev. 2009;46(5):603-18. doi: 10.1682/jrrd.2007.03.0052. PMID 19882494